CLINICAL TRIAL: NCT05185648
Title: Analysis of Current Situation and Evaluation of Trauma Treatment Training in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2021-0675
Record Dates: First submitted 2021-12-06; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-07

CONDITIONS: Train Accident Involving Explosion, Passenger Injured; Train Collision With Streetcar, Pedestrian Injured; Trauma Injury; Train Accident Involving Burning, Passenger Injured
Keywords: trauma training; trauma care
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- post-training scores (Experimental): evaluating qualities of trauma care after standard trauma traning
  Interventions: Behavioral: standard trauma care taining

INTERVENTIONS:
Behavioral: standard trauma care taining — trauma care training

SUMMARY:
This study will rely on the training course of CTCT project to conduct standardized training for trauma practitioners in China. And the quality of training will be stratified research; Continuously improve the quality of trauma treatment and improve the prognosis of trauma patients.

ELIGIBILITY:
All CTCT participants from different administrative districts of China registered for standardized and procedural CTCT curriculum . All trainees have finished the general survey of personal background, trauma care status in local hospitals and pre-training tests of trauma knowledge. After CTCT curriculum and hifidelity trauma simulation training, they were also needed to finish post-training test about the initial evaluation of various kinds of traumas. The pre- and post-training examination were constantly about trauma evaluation of major trauma patients.

Inclusion criteria: Trainees who attended on CTCT curriculum. Exclusion criteria: Rejection for supplying training information, in-completed CTCT training information, lack of pre- and/or post-training scores.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
training scores | Day 1.5
  Commare between pre- and post-training scores

SECONDARY OUTCOMES:
score difference | Day 1.5
  evaluation the improvement of trauma care

CONTACTS AND LOCATIONS:
Overall Officials: yongan xu, doctor, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University